CLINICAL TRIAL: NCT00000808
Title: A Phase I Study of Safety and Pharmacokinetics of Nevirapine in HIV-1 Infected Pregnant Women and Neonates Born to HIV-1 Infected Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 250; 11227 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Nevirapine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
To determine the bioavailability, pharmacokinetics, and short-term safety and tolerance of nevirapine in HIV-1 infected pregnant women and their newborns when nevirapine is given to the mother during active labor, and when their neonates are dosed during the first week of life. To determine the short-term safety profile of mothers receiving zidovudine (AZT) who received nevirapine during active labor, and their neonates who received no dose, a single dose, or multiple doses of nevirapine and who are receiving AZT during the first 6 weeks of life.

Treatment of HIV-1 infected pregnant women during active labor may result in therapeutic levels of nevirapine in the neonate at the time of exposure to HIV-1 during parturition, decreasing the neonate's risk of infection.

DETAILED DESCRIPTION:
Treatment of HIV-1 infected pregnant women during active labor may result in therapeutic levels of nevirapine in the neonate at the time of exposure to HIV-1 during parturition, decreasing the neonate's risk of infection.

Pregnant women in active labor receive single doses of oral nevirapine. The neonates of the first 4-6 (PER AMENDMENT 8/27/96, was 4) mothers receive no drug, while the neonates of the second 4-6 (PER AMENDMENT 8/27/96, was 4) patient cohort receive a single dose of nevirapine. If neonatal antiviral levels of nevirapine are not sustained for 7 days after the single dose, a third cohort of 4-6 (PER AMENDMENT 8/27/96, was 4) pregnant women will receive a single dose of nevirapine and their neonates will receive multiple doses of nevirapine to maintain an antiviral effect for 7 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT (mothers and neonates).
* Oral asthma inhalers (mothers).

Concurrent Treatment:

Allowed:

* Phototherapy (neonates).

MOTHERS must have:

* HIV infection.
* Estimated gestational age >= 34 weeks.
* No active opportunistic infection at study entry.

PER AMENDMENT 8/27/96:

* A pre-enrollment plasma HIV-1 RNA level greater than 10,000 copies/ml.

Exclusion Criteria

Co-existing Condition:

MOTHERS with the following symptoms or conditions are excluded:

* Intrauterine growth retardation.
* Fetal anomaly incompatible with life as determined by pre-entry ultrasound.
* Participation during current pregnancy in any other therapeutic or vaccine perinatal trial.
* Known hypersensitivity to any benzodiazepine.
* Serious bacterial infection.

Concurrent Medication:

Excluded:

* Any antiretroviral other than AZT.
* Corticosteroids (other than oral asthma inhalers).
* Anticoagulants.
* Any clavulanic acid-containing formulation (e.g., Augmentin, Timentin).
* Benzodiazepines other than study drug.
* Phenobarbital.
* Barbiturates.
* Antacids.
* Magnesium sulfate.

Prior Medication:

Excluded:

* Prior nevirapine.

Current use of illicit substances and/or active chronic alcohol use.

Ages: 13 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49
Dates: Study Completion 1998-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sullivan JL, Study Chair; Sperling R, Study Chair
Locations (16):
- United States (15):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Connecticut Children's Med Ctr - Pediatric, Hartford, Connecticut
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Vazquez E. Two bucks a baby. Posit Aware. 1997 Mar-Apr;8(2):15. PMID 11364450
- [Background] Benson M, Shannon M. Nevirapine: ethical dilemmas and care for HIV-infected mothers. Focus. 1995 Jun;10(7):5-6. PMID 11362587
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] Mirochnick M, Sullivan J, Cort S, Mcnamara J, Fenton T, Sperling R. Safety and pharmacokinetics (pk) of nevirapine (NVP) in HIV-I infected pregnant women and their newborns. ACTG Protocol 250 Team. American Pediatric Association and Society for Pediatric Research annual meeting; 1996 May 6-10; Washington, D.C. Pediatr AIDS HIV Infect. 1996 Aug;7(4):280 (unnumbered abstract)
- [Background] Mirochnick M, Fenton T, Gagnier P, Pav J, Gwynne M, Siminski S, Sperling RS, Beckerman K, Jimenez E, Yogev R, Spector SA, Sullivan JL. Pharmacokinetics of nevirapine in human immunodeficiency virus type 1-infected pregnant women and their neonates. Pediatric AIDS Clinical Trials Group Protocol 250 Team. J Infect Dis. 1998 Aug;178(2):368-74. doi: 10.1086/515641. PMID 9697716